CLINICAL TRIAL: NCT04712838
Title: Study on the Bioavailability of SHR0302 Tablets With 3 Different Formulations in Healthy Subjects (Single Center, Random, Open, 3 Cycles, 6 Sequences)
Brief Title: Study on the Bioavailability of SHR0302 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SHR0302-108
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ivarmacitinib

STUDY DESIGN:
Intervention Model Description: The relative bioavailability of SHR0302 tablets with three different formulations
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- group A (Experimental)
  Interventions: Drug: SHR0302
- group B (Experimental)
  Interventions: Drug: SHR0302
- group C (Experimental)
  Interventions: Drug: SHR0302
- group D (Experimental)
  Interventions: Drug: SHR0302
- group E (Experimental)
  Interventions: Drug: SHR0302
- group F (Experimental)
  Interventions: Drug: SHR0302

INTERVENTIONS:
Drug: SHR0302 — Group A subjects were given oral F1 、F2 and F3 version SHR0302
  Arms: group A
Drug: SHR0302 — Group B subjects were given oral F1 、F3 and F2 version SHR0302
  Arms: group B
Drug: SHR0302 — Group C subjects were given oral F2 、F1 and F3 version SHR0302
  Arms: group C
Drug: SHR0302 — Group D subjects were given oral F2 、F3 and F1 version SHR0302
  Arms: group D
Drug: SHR0302 — Group E subjects were given oral F3 、F1 and F2 version SHR0302
  Arms: group E
Drug: SHR0302 — Group F subjects were given oral F3 、F2 and F1 version SHR0302
  Arms: group F

SUMMARY:
The study is being conducted to evaluate the safety, and the relative bioavailability of SHR0302 tablets with three different formulations in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to sign an informed consent form before the start of the relevant activities of this trial, understand the procedures and methods of this trial, and be willing to strictly abide by the clinical trial protocol to complete this trial
2. 18~45 years old (including both ends, subject to when signing the informed consent form), healthy male
3. Weight ≥ 50 kg, and body mass index (BMI): 19~26 kg/m2 (including both ends)
4. Those who have signed the informed consent and have no birth plan within 6 months after the last administration, and agree to take effective contraceptive measures
5. Able to communicate well with the researcher, and understand and comply with the requirements of this research

Exclusion Criteria:

1. Suspected of being allergic to the study drug or any ingredient in the study drug, or allergic
2. Those who have participated in clinical trials of any drugs and medical devices within six months before screening (subject to the signed informed consent form)
3. Subjects with any systemic inflammatory disease or autoimmune disease
4. Subjects with a history of recurrent herpes zoster, disseminated herpes zoster or disseminated herpes simplex
5. Subjects with a history of malignant tumors
6. Subjects with mental or neurological diseases, unwilling to communicate or have language barriers, unable to fully understand and cooperate
7. Those who have a history of tuberculosis (TB) within six months before screening, or have clinical or imaging evidence of active or occult TB
8. Routine blood examination during the screening period: white blood cell count <3.0×109/L and/or neutrophil count <1.5×109/L
9. Subjects Those with serum creatinine> 1.5 mg/dL (133 μmol/L) at the time of screening
10. At the time of screening, 12-ECG check QTcF>450 ms or there are other abnormal conditions judged by the investigator to be clinically meaningful
11. Those who are positive for hepatitis B surface antigen, hepatitis C antibodies, syphilis antibodies, and HIV antibodies
12. Those who smoked more than 5 cigarettes daily in the 3 months before screening and cannot stop using any Tobacco products
13. Those who drink regularly in the 6 months before screening, drink more than 14 units of alcohol per week (1 unit = 285 mL of beer, 25 mL of spirits, or 100 mL of wine) and cannot stop using any alcoholic products during the trial; those who have a positive alcohol breath test
14. People who have a history of drug abuse, drug dependence or a positive urine drug abuse screening before administration, including: morphine, methamphetamine (methamphetamine), ketamine, cocaine, ecstasy (dimethylene) Dioxyamphetamine), cannabis (tetrahydrocannabinolic acid)
15. Those who have had any surgery within 6 months before screening
16. Infections that require antimicrobial (virus, bacterial, fungal, and parasitic infections) treatment that occurred within 4 weeks before screening
17. Donated blood (or blood loss) within 3 months before screening and donated blood (or blood loss) ≥400 mL, or received blood transfusion
18. Those who have had any acute disease that has been determined by the investigator to be clinically significant within 1 month before screening
19. Those who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products within 14 days before taking the study drugs; those who plan to take non-study drugs or health products during the trial period
20. The 48 hours before the first dose until the end of the study, the subject refused to stop any methyl yellow Purine beverages or foods, such as coffee, tea, cola, chocolate, etc.; The 7 days before the first dose until the end of the study, the subject refused to stop using any beverages or foods containing grapefruit; there are special dietary requirements that cannot be consistent Eaters
21. Physical examination, vital signs, laboratory examinations, chest X-ray or chest CT, abdominal ultrasound and other abnormal and clinically meaningful examination results
22. The researcher believes that there are other subjects who are not suitable for participating in the research

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
The peak plasma concentration (Cmax) of SHR0302. | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose.
  Based on the PK concentration data set, calculate the peak plasma concentration of SHR0302 by non-compartmental analysis.
Area Under the Plasma Concentration Versus Time Curve (AUC) of SHR0302. | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose.
  Based on the SHR0302 plasma concentration data set, calculate the Area Under the Plasma Concentration Versus Time Curve of SHR0302 by non-compartmental analysis.
The relative bioavailability of SHR0302 tablets with 3 different formulations. | through study completion, an average of 1 month.
  The mixed effect model is used to estimate the least square mean difference and 90% confidence interval between different formulations, and then take the antilog to obtain the estimate of the ratio of the least square geometric mean of the corresponding PK parameter and the 90% confidence interval Time.

SECONDARY OUTCOMES:
The Peak Time (Tmax) of SHR0302. | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose.
  Based on the SHR0302 plasma concentration data set, calculate the time to reach peak plasma concentration of SHR0302 by non-compartmental analysis.
The Elimination half-life (T1/2) of SHR0302. | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose.
  Based on the SHR0302 plasma concentration data set, calculate the time required for the blood concentration of SHR0302 to drop by half.
The Clearance (CL/F) of SHR0302. | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose.
  Based on the SHR0302 plasma concentration data set, calculate the clearance of SHR0302 by non-compartmental analysis.
The apparent volume of distribution (Vz/F) of SHR0302. | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post-dose.
  Based on the SHR0302 plasma concentration data set, calculate the apparent volume of distribution of SHR0302 by non-compartmental analysis.
Incidence of adverse events. | through study completion, an average of 1 month
  laboratory abnormalities (based on hematology, biochemistry, coagulation function, and urinalysis tests), vital sign measurements (include blood pressure, pulse rate, respiratory rate, and body temperature) and 12-Lead electrocardiogram.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Beijing,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided